CLINICAL TRIAL: NCT01120119
Title: Clinical Study to Evaluate the Efficacy of 1,25(OH)2D3 (Calcitriol) Versus Placebo in Recent Onset Type 1 Diabetes(IMDIAB XIII)
Brief Title: Efficacy of Calcitriol in Recent Onset Type 1 Diabetes
Acronym: IMDIABXIII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Paolo Pozzilli/Principal Investigator, University Campus Bio Medico
Other Study IDs: CLF-1 2005-000751-15
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2005-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcitriol (Experimental)
  Interventions: Drug: Calcitriol
- placebo (Placebo Comparator)
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol

SUMMARY:
Reduction in vitamin D levels has been reported in subjects with recent onset type 1 diabetes. Several studies suggest that vitamin D supplementation in early childhood decreases the risk of developing type 1 diabetes, therefore vitamin D deficiency might play a role in the disease pathogenesis. We investigated whether the supplementation of the active form of vitamin D (calcitriol) in subjects with recent-onset type 1 diabetes can protect residual beta cell function evaluated by C peptide and improve glycaemic control as evaluated by HbA1c and insulin requirement.

Thirty-four subjects (age range 11-35 years, median 18 years) with recent-onset type 1 diabetes (<12 weeks duration) and high basal C-peptide >0.25 nmol/l were randomized in a double-blind trial to calcitriol (the active form of vitamin D, 1.25-dihydroxyvitamin D3 [1,25-(OH)2D3] ) at the dose of 0.25 ug/day or placebo, and followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of type 1 diabetes according to the American Diabetes Association (ADA) guidelines;
2. age at presentation between 11 and 35 years;
3. duration of clinical disease (since the beginning of insulin therapy) <12 weeks;
4. baseline C-peptide >0.25 nmol/l;
5. no medical contra-indications or any other major chronic disease;
6. willingness and capability to participate in a regular follow-up.

Exclusion Criteria:

1. cardiovascular disease;
2. renal disease;
3. liver disease;
4. neurological disorders;
5. allergic diathesis;
6. hyperparathyroidism;
7. neoplasia.

Ages: 11 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

PRIMARY OUTCOMES:
C peptide
  evaluation of baseline and stimulated C peptide

SECONDARY OUTCOMES:
Glycometabolic control
  To measure insulin requirement and HbA1c

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - University Campus Bio Medico, Rome
  - Bambino Gesù Children's Hospital, Rome
  - Catholic University,, Rome
  - Sandro Pertini Hospital, Rome
  - University Sapienza, Rome

REFERENCES:
- [Background] Pitocco D, Crino A, Di Stasio E, Manfrini S, Guglielmi C, Spera S, Anguissola GB, Visalli N, Suraci C, Matteoli MC, Patera IP, Cavallo MG, Bizzarri C, Pozzilli P; IMDIAB Group. The effects of calcitriol and nicotinamide on residual pancreatic beta-cell function in patients with recent-onset Type 1 diabetes (IMDIAB XI). Diabet Med. 2006 Aug;23(8):920-3. doi: 10.1111/j.1464-5491.2006.01921.x. PMID 16911633
- [Derived] Bizzarri C, Pitocco D, Napoli N, Di Stasio E, Maggi D, Manfrini S, Suraci C, Cavallo MG, Cappa M, Ghirlanda G, Pozzilli P; IMDIAB Group. No protective effect of calcitriol on beta-cell function in recent-onset type 1 diabetes: the IMDIAB XIII trial. Diabetes Care. 2010 Sep;33(9):1962-3. doi: 10.2337/dc10-0814. PMID 20805274